CLINICAL TRIAL: NCT05952583
Title: Selective Fetal Growth Restriction in Monochorionic Twins - an International Investigation
Acronym: CONTRAST
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Karolinska University Hospital (Other); BCNatal Fetal Medicine Research Center (Unknown); MOUNT SINAI HOSPITAL (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, ejtverweij, Principal Investigator, Leiden University Medical Center
Other Study IDs: CONTR
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Twin; Pregnancy, Affecting Fetus or Newborn; Fetal Growth Retardation; Twin Monochorionic Diamniotic Placenta; Twin Diseases
Keywords: sFGR; sIUGR; selective fetal growth restriction
MeSH Terms: conditions — Fetal Growth Retardation; Diseases in Twins | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sFGR cohort: Monochorionic diamniotic twin pregnancies complicated by sFGR (diagnosed before 28 weeks of gestational age)
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Additional ultrasound measurements during pregnancy

SUMMARY:
Optimal diagnostic management and underlying pathophysiological mechanisms of selective fetal growth restriction (sFGR) in monochorionic diamniotic (MCDA) twin pregnancies have not been fully clarified.

The current diagnostic classification system based on three different umbilical artery flow patterns has no increasing scale of severity and the predictive value is limited. Since there is no treatment available for sFGR, predicting fetal deterioration is key in preventing single or double fetal demise. Outcome prediction is furthermore important in the selection of cases that will be offered selective reduction (to provide the larger twin with better prospects), as well as determining monitor frequency and possible hospital admission. As outcome prediction is clinically challenging, patient counselling is too, and parents often encounter a great deal of uncertainty during the pregnancy.

Furthermore, little is known about the brain development of sFGR children (both during pregnancy and after birth). Moreover, the psychological impact of an sFGR pregnancy of the future parent)s) has not been studied before. The impact of these factors should be taken into account during patient counseling, which is currently not the case.

By our knowledge, this is the first international, multicenter, prospective cohort study on that will address the abovementioned questions and knowledge gaps in MCDA pregnancies complicated by selective fetal growth restriction.

DETAILED DESCRIPTION:
Selective fetal growth restriction (sFGR) in monochorionic twins may negatively impact the pregnancy. There is a substantial risk of fetal deterioration resulting in (iatrogenic) preterm birth or even intrauterine demise of one, or both fetuses. There are important unresolved challenges on a diagnostic level and underlying pathophysiological mechanisms of sFGR have not been fully clarified.

The current diagnostic classification system based on three different umbilical artery flow patterns has no increasing scale of severity and the observed flow patterns may be volatile in nature. This hinders optimal diagnostic management and complicates outcome prediction as the survival outcome differs per umbilical artery flow type. Consequently, parents encounter a great deal of uncertainty during the pregnancy. Since there is no treatment available for sFGR, predicting fetal deterioration is key in preventing single or double demise.

By testing several predictors, the investigators are aiming to improve outcome prediction at the time of sFGR diagnosis. The investigators furthermore hypothesize that additional ultrasound parameters could be of benefit in making the current classification system more accurate and less variable. Extensive histological placental examinations will shine a light on microscopic abnormalities which can increase our knowledge of the pathophysiology. Examining neurodevelopment of sFGR twins at two years of age will additionally be of great value for our understanding of the impact of sFGR and contribute to adequate patient counselling. Our study will evaluate the impact of a sFGR pregnancy on parental mental health and parent-to-infant(s) attachment, which has not been carried out this extensively before.

ELIGIBILITY:
Inclusion Criteria:

* MCDA twin pregnancy
* Diagnosis of sFGR before 28+0 weeks of GA (independent of Doppler flows)
* Pregnant woman ≥ 18 years and able to consent
* Partner (who has (future) parental responsibility - if applicable) ≥ 18 years and able to consent
* Written informed consent of both parents (if applicable) for participation in the longitudinal follow-up until 2 years after birth)

Exclusion Criteria:

* The presence of lethal anomalies (one or both fetuses)
* Multiple pregnancy higher order than twins;
* TTTS/TAPS present at moment of sFGR diagnosis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MCDA pregnancies complicated by sFGR pregnancies that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | 2 years
  The composite outcome consists of fetal single or double demise, including selective fetal reduction and/or an iatrogenic elective birth < 32 weeks of gestational age because of fetal distress).

SECONDARY OUTCOMES:
Ultrasound parameters | 2 years
  Explanatory analysis of ultrasound parameters over course of sFGR pregnancy
Prenatal and postnatal attachment | 2 years
Post-traumatic stress | 2 years
PARCA-R evaluation | 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Leiden University Medical Center, Leiden, South Holland, Netherlands
- BCNatal, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.foetaletherapie.nl/contrast-studie